CLINICAL TRIAL: NCT06353828
Title: A Phase 2a, Randomized, Double-blind, Placebo Controlled Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of IcBD-01 Enema for the Treatment of Active Ulcerative Colitis
Brief Title: Phase 2a Study to Evaluate IcBD-01 Enema in Active Ulcerative Colitis Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CannaMore Biotechs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICBD-UC-01
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IcBD-01 (Experimental): IcBD-01 is a novel Cannabidiol enema formulation
  Interventions: Drug: CBD, synthetic form
- placebo (Placebo Comparator): placebo enema formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD, synthetic form — Cannabidiol enema
  Arms: IcBD-01
Drug: Placebo — placebo enema
  Arms: placebo

SUMMARY:
Ulcerative proctitis can lead to considerable morbidity, and the available treatment options are limited. Cannabidiol (CBD), a non-psychotropic ingredient of Cannabis sativa, possesses potent immunomodulatory and anti-inflammatory properties as described in both acute and chronic animal models of inflammation, including IBD models.

Based on positive safety and initial efficacy profiles of CBD found in IBD animal and clinical studies, the main aim of this study is to evaluate the safety, tolerability and efficacy of a novel enema formulation of CBD for the treatment of active ulcerative proctitis.

DETAILED DESCRIPTION:
This study consists of 2 stages:

Stage 1. Feasibility - Open label stage:

Up to fourteen patients will be enrolled in this stage and receive a CBD enema formulation for 12 weeks treatment period.

If results of this stage prove to be safe and with clinical effect (reduction of 3 points in full Mayo score in at least 50% of patients), the study will proceed to stage 2.

Stage 2. Randomized, placebo controlled blinded stage:

Subjects will be randomized in a 2:1 ratio and receive the drug/placebo enema for a 12 weeks treatment period.

Patients will be assessed for full Mayo score on visit 1 and week 12, and partial Mayo score every visit. Patients will assessed by a clinician using the self reported outcome (PRO) scale every visit. Sigmoidoscopy will be performed at baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of UC at least 3 months prior to the Screening Visit
3. Patients who were not treated rectally for UC in the last 3 days.
4. UC patients with active disease and being treated with stable doses of biologics (at least 2 months), and/or steroids (at least 1 months) and/or oral mesalazine (at least 2 months at stable dose (4 gr)) or non-treated patients)
5. Full Mayo score ≥4 to < 9 (range: 0-12) prior to enrolment in the study
6. Patients that did not respond to Mesalamine treatment.
7. Non-pregnant (via negative pregnancy test)/non-breast-feeding women and women with no intention to become pregnant/to breast-feed during the term of the trial and for at least one month after cessation of IcBD-01 treatment
8. Male subject with female partner(s) of child-bearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for one month after final IMP administration.
9. Subject able to provide written informed consent
10. Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Diagnosis of severe extensive pancolitis
2. Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis, or diverticular disease-associated colitis
3. Complete resection of the colon with the need of a pouch
4. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis, atypical mycobacterial disease, and herpes zoster), human immunodeficiency virus (HIV), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) or oral antibiotics within 4 weeks of screening
5. Sexual transmitted diseases
6. Using rectal formulations (such as Mesalazine) for the last 3 days
7. Subjects who have received any investigational drug or used investigational device in the last 2 months
8. Serious psychiatric or psychological disorders
9. Active consumption of illicit drugs including cannabis or derivatives for at least 1 months prior to the study
10. Patients with short bowel syndrome, symptomatic stricture, abscess, recent history (within the previous 3 months) of abdominal surgery
11. Patients with significant cardiac, hepatic, respiratory disease comorbidities or active malignancy
12. Renal comorbidity: eGFR< 30 mL/min/1.73 m2 (note: CKD Grade 4 is defined as eGFR 15-29 mL/min/1.73 m2)
13. Patient who is taking immunomodulatory medications for other indication(s)
14. Women of child-bearing potential who intend to become pregnant or who are pregnant or breastfeeding or male subjects with female partners who intend to get pregnant or breastfeed during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Full Mayo Score | 12 weeks
  The Mayo Score is used to assess the severity of ulcerative colitis and can range from 0-12, with higher scores indicating worse severity.

SECONDARY OUTCOMES:
Change in Partial Mayo Score | 12 weeks
  The partial Mayo Score is used to assess the severity of UC and does not include the endoscopic parameter. Can range from 0-9, with higher scores indicating worse severity.
Change in patient reported outcome (PRO-UC) | 12 weeks
  PRO-UC Diary is a tool to quantify the patient perspective in terms of how they feel and function. Can range from 0-20, with higher scores indicating worse severity
Change in endoscopic Mayo subscore in distal 15 cm of anus | 12 weeks
  Efficacy will be determined through the use of the Mayo Endoscopic Subscore.
Change in the length of the inflamed colon | 12 weeks
  Length of inflamed colon (Mayo subscore) will be measured through endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No